CLINICAL TRIAL: NCT00132769
Title: A Randomized, Placebo-Controlled, Parallel-Group, Double-Blind, 12-Week Study to Assess the Clinical Efficacy, Safety, and Tolerability of MK-0873 in Rheumatoid Arthritis
Brief Title: A Study of a Novel Investigational Drug in Rheumatoid Arthritis Patients (MK-0873-012)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0873-012; 2005_029 (Other: Telerex Study Number)
Record Dates: First submitted 2005-08-02; First posted 2005-08-22 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — MK 0873

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-0873 (Experimental): MK-0873 1.25 mg twice daily for 12 weeks
  Interventions: Drug: MK-0873
- Placebo (Placebo Comparator): Matching placebo to MK-0873 1.25 mg twice daily for 12 weeks
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK-0873 — MK-0873 1.25 mg twice daily for 12 weeks
  Arms: MK-0873
Drug: Comparator: Placebo — Matching placebo to MK-0873 1.25 mg twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
This study will look at whether this new drug is effective in the treatment of rheumatoid arthritis, and at whether it is safe and well-tolerated by participants with the disease.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis, according to the American College of Rheumatology criteria, with active disease despite current medications
* Other criteria also apply

Exclusion Criteria:

* Other major illnesses
* Past history of certain other disorders
* Certain prohibited medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-0873: Participants receive MK-0873 1.25 mg twice daily for 12 weeks
- Placebo: Participants receive matching placebo to MK-0873 twice daily for 12 weeks
Period: Overall Study
Arm/Group | MK-0873 | Placebo
Started | 53 | 53
Completed | 42 | 42
Not Completed | 11 | 11
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lack of Efficacy | 7 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0873 | Placebo | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (9.30) | 53.5 (8.99) | 52.3 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 75
  Male | 18 | 13 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Swollen Joint Count
Description: Swollen joint count (SJC) was determined by assessing 66 joints (33 right side, 33 left side) for swelling using the following grading system: 0=Absent, 1=Detectable synovial thickening without loss of bony contours, 2=Loss of distinctiveness of bony contours, or 3=Bulging synovial proliferation with cystic characteristics. The total number of joints graded 1, 2, or 3 were then counted to yield the SJC. SJC ranged from 1-66, with increasing score indicating greater number of swollen joints. SJC was averaged over weeks 8, 10 and 12 to yield a Treatment Period Mean. Change from Baseline = Treatment Period Mean SJC - Baseline SJC.
Time Frame: Baseline and the average of Treatment Weeks 8, 10 and 12
Population: The All Patients Treated (APT) population consisted of all participants with a baseline and at least one postbaseline observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 53 | 53
score on a scale | -7.20 [-9.54 to -4.86] | -8.68 [-10.97 to -6.39]
Statistical Analysis 1: Comparison: MK-0873 vs Placebo; Test type: Superiority or Other; p = 0.278, ANCOVA; Difference in LS Mean = 1.48, 95% CI 2-sided [-1.21 to 4.18]

2. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% Response [ACR20]
Description: Participants were categorized as meeting ACR20 criteria when they had at least 20% improvement from Baseline in tender and swollen joint counts, and improvement from Baseline in at least 3 of 5 of the following domains: Pain Visual Analog Scale (VAS), Patient Global Assessement, Physician Global Assessment, Patient Physical Function (Disability) Score and acute-phase reactant (Erythrocyte Sedimentation Rate [ESR] or C-Reactive Protein [CRP]). The average percentage of participants that met the ACR20 responder criteria over Treatment Weeks 8, 10 and 12 was calculated.
Time Frame: Baseline and the average of Treatment Weeks 8, 10 and 12
Population: The APT population consisted of all participants with a baseline and at least one postbaseline observation.
Measure: Number; unit: percentage of participants
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 53 | 53
percentage of participants | 39.62 | 45.28
Statistical Analysis 1: Comparison: MK-0873 vs Placebo; Test type: Superiority or Other; p = 0.543, Cochran-Mantel-Haenszel; Difference in Percent = -5.66, 95% CI 2-sided [-24.45 to 13.13]

3. Secondary Outcome: Change From Baseline in Tender Joint Count
Description: Tender joint count (TJC) was to be determined by assessing 68 joints (34 right side, 34 left side) for pain using the following grading system: 0=No pain, 1=Patient states that there is pain, 2=Patient states that there is pain and winces, or 3=Patient states that there is pain, winces, and withdraws. The total number of joints graded 1, 2, or 3 were then to be counted to yield the TJC. TJC ranges from 1-68, with increasing score indicating greater number of tender joints. TJC was to be averaged over weeks 8, 10, and 12 to yield a Treatment Period Mean. Change from Baseline = Treatment Period Mean TJC - Baseline TJC.
Time Frame: Baseline and the average of Treatment Weeks 8, 10 and 12
Population: No additional analyses were performed if the primary (Swollen Joint Count) and major secondary (ACR20) outcome measures resulted in a p-value of >0.05.
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Patient Global Assessment of Disease Activity
Description: At each clinic visit, participants were to assess disease activity using a 100 mm visual analog scale (VAS) in reponse to the question: "Considering all the ways your arthritis affects you, mark an (X) through the line for how well you are doing." The VAS ranges from "Very Well" (0) to "Very Poor" (100). The mean score at Treatment Weeks 8, 10 and 12 was calculated. A lower score indicates a better disease activity.
Time Frame: The average of Treatment Weeks 8, 10 and 12
Population: as for outcome 3
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Investigator Global Assessment of Disease Activity
Description: At each clinic visit, the Investigator was to make a global assessment of participant disease activity on a 5-point Likert scale with grading as follows: 1=Very well, 2=Well, 3=Fair, 4=Poor, or 5=Very poor (scale range: 1-5). A lower score indicates a more positive assessment of participant disease activity.
Time Frame: Treatment Week 12
Population: as for outcome 3
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Global Assessment of Response to Therapy
Description: Participants were to rate their overall response to the study drug on a 5-point Likert scale with grading as follows: 0=None, 1=Poor, 2=Fair, 3=Good, or 4=Excellent (scale range: 0-4). A higher score indicates a more positive response to study drug.
Time Frame: Treatment Week 12
Population: as for outcome 3
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Health Assessment Questionnaire Disability Index
Description: The Stanford Health Assessment Questionnaire Disability Index assesses participant functional ability based on 20 questions in 8 categories of functioning: dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Responses range from 0=No disability to 3=Completely disabled. The score for each category subscale is the single response within the category with the highest score (greatest difficulty). The overall score for the Disability Index is the mean of the 8 category scores and also ranges from 0-3, with a lower score indicating less disability.
Time Frame: The average of Treatment Weeks 8, 10 and 12
Population: as for outcome 3
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patient's Assessment of Pain
Description: At each clinic visit, participants were to assess their amount of pain due to arthritis during the previous 48 hours on a 100 mm visual analog scale (VAS) that ranged from "No pain" (0) to "Extreme pain" (100). A lower score indicates less pain.
Time Frame: Treatment Week 12
Population: as for outcome 3
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Ratio of On-treatment C-Reactive Protein to Baseline C-Reactive Protein
Description: C-reactive protein levels rise in response to inflammation in the body. The ratio of On-treatment serum C-reative protein:Baseline serum C-reactive protein was calculated to determine a treatment effect. On-treatment C-reactive protein = the mean of serum C-reactive protein levels for Treatment Weeks 8, 10 and 12. A ratio of less than 1.0 is consistent with lower inflammation and was to be considered an improvement.
Time Frame: Baseline and the average of Treatment Weeks 8, 10 and 12
Population: The APT population consisted of all participants with a baseline and at least one postbaseline observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | MK-0873 | Placebo
Number analyzed (Participants) | 53 | 53
ratio | 0.90 [0.70 to 1.16] | 1.08 [0.85 to 1.38]
Statistical Analysis 1: Comparison: MK-0873 vs Placebo; Test type: Superiority or Other; p = 0.225, ANCOVA; LS mean ratio between treatments = 0.84, 95% CI 2-sided [0.63 to 1.12]

ADVERSE EVENTS:
Time Frame: Up to 4 weeks
Description: The safety population consisted of all participants who took at least one dose of study drug.
Arm/Group | MK-0873 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/53 | 2/53
Other Adverse Events (participants affected / at risk) | 10/53 | 4/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0873 (N=53) | Placebo (N=53)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mental Disorder (Psychiatric disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-0873 (N=53) | Placebo (N=53)
Diarrhoea (Gastrointestinal disorders) | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.